CLINICAL TRIAL: NCT04770701
Title: Extracts of Plants Eclipta Prostrata, Dioscorea Cirrhosa, Phyllanthus Urinaria, Adenosma Glutinosum, Impatiens Balsamina and Ascorbic Acid Use for in Protecting and Increasing CD4+ T Lymphocytes; B Lymphocytes Level in HIV/AIDS Patients.
Brief Title: Protect and Improve Cluster of Differentiation 4 (CD4) Cells and B Cells Lymphocytes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Trieu, Nguyen Thi, M.D. (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HIV / AIDS
Record Dates: First submitted 2021-01-03; First posted 2021-02-25 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: HIV-1-infection; AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — A1A0 ATPase, Methanosarcina mazei

STUDY DESIGN:
Intervention Model Description: 60 people were recruited HIV / AIDS positive between the ages of 20 and 60 and divided into 2 groups according to a random distribution.
Who Masked: Outcomes Assessor
Masking Description: The group of HIV / AIDS uses drugs under study. The group of HIV / AIDS uses a placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ahah drug (Experimental): Participants have a decline in CD4 + T-lymphocytes is the hallmark of the human immunodeficiency virus (HIV)-1 infection.
  Characterized by rapid loss of resistance: AIDS
  * Dermatitis, mouth ulcers, skin rash, itching, weight loss
  * Hepatitis C virus (HCV) (+), Hepatitis B virus (HBV) (+), Tuberculosis (+)
  Ahah composition contains the following ingredients (concentrated extracts of plants):
  Eclipta prostrata 200mg, dioscorea cirrhosa 200mg, phyllanthus urinaria 150mg, adenosma glutinosum 150mg, impatiens balsamina 75mg and ascorbic acid 250mg
  Interventions: Drug: Ahah Drug
- Ahah Placebo (Experimental): Participants have a decline in CD4 + T-lymphocytes is the hallmark of the human immunodeficiency virus (HIV)-1 infection.
  Characterized by rapid loss of resistance: AIDS
  * Dermatitis, mouth ulcers, skin rash, itching, weight loss
  * Hepatitis C virus (HCV)(+), Hepatitis B virus (HBV)(+), Tuberculosis (+)
  Ahah composition placebo (Ahah not containing concentrated extracts of plants Eclipta prostrata 200mg, dioscorea cirrhosa 200mg, phyllanthus urinaria 150mg, adenosma glutinosum 150mg, impatiens balsamina 75mg and ascorbic acid 250mg)
  Interventions: Device: Ahah Placebo

INTERVENTIONS:
Drug: Ahah Drug — - Composition Ahah containing concentrated extracts of plants: Eclipta prostrata 200mg, dioscorea cirrhosa 200mg, phyllanthus urinaria 150mg, adenosma glutinosum 150mg, impatiens balsamina 75mg and ascorbic acid 250mg
  -Take 1tablet x 2 times / 24 hours. Maintained for 9 months.
  Other Names: Ahah
  Arms: Ahah drug
Device: Ahah Placebo — - Composition Ahah (not containing concentrated extracts of plants): Eclipta prostrata 200mg, dioscorea cirrhosa 200mg, phyllanthus urinaria 150mg, adenosma glutinosum 150mg, impatiens balsamina 75mg and ascorbic acid 250mg)
  -Take 1tablet x 2 times / 24 hours. Maintained for 9 months.
  Other Names: Ahah
  Arms: Ahah Placebo

SUMMARY:
This is a plant-based medication used to increase the amount, protect, and reduce HIV's impact on T and B lymphocytes.

DETAILED DESCRIPTION:
Dioscorea cirrhosa, impatiens balsamina, eclipta prostrata, phyllanthus urinaria, adenosma glutinosum, and ascorbic acid are used to elevate T and B lymphocytes level, protect their cells membrane, decrease the damage of HIV on CD4+ T.

In detail, Diosgenin presented in dioscorea cirrhosa is a precursor of cortisol. Dioscorea cirrhosa when combined with ascorbic acid helps to balance cortisol levels which reduces cell inflammation. Flavonoids of dioscorea cirrhosa also help to increase CD4+ T levels.

impatiens balsamina can be used as an antitoxin alternative against bacteria or viruses. Flavonoids in impatiens balsamina, such as kaempferol, quercetin, rutin, astragalin, have the ability to reduce the virus's impact on T lymphocyte, protect their cell membrane, produce antihistamine, protect the cell from inflammation.

Targeted flavonoids in eclipta prostrata, phyllanthus urinaria, adenosma glutinosum are used to cell repair, protect and increase CD4+ T production.

Ascorbic acid in combination with herbal extracts creates a favorable environment for body metabolism, improves the medication's effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Participants have a decline in CD4 + T-lymphocytes is the hallmark of HIV-1 infection.

Characterized by rapid loss of resistance: AIDS

* Dermatitis, mouth ulcers, skin rash, itching, weight loss
* HCV (+), HBV (+), Tuberculosis (+)

Exclusion Criteria:

* Cancer under all form

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2021-01-08 (Actual); Study Completion 2021-01-10 (Actual)

PRIMARY OUTCOMES:
The CD4 cell count measurement | - 9 months
  HIV is a fatal infection, characterized by the targeting and destruction of CD4 T lymphocytes in the peripheral blood.

CONTACTS AND LOCATIONS:
Overall Officials: Tran Minh Duc, Dr., Principal Investigator — Trieu, Nguyen Thi, M.D.
Locations (2):
- Saigon Biopharma LLC, Wilmington, Delaware, United States
- Saigon Biopharma Company Limited, Ho Chi Minh City, Vietnam